CLINICAL TRIAL: NCT05100693
Title: Non-invasive Removal of the Smart Tracheal Occlusion Device for Fetal Congenital Diaphragmatic Hernia: A Feasibility Study
Brief Title: Smart Removal for Congenital Diaphragmatic Hernia
Acronym: SmartRemoval
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Jan Deprest, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S65423
Record Dates: First submitted 2021-09-20; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedure FETO with the Smart-TO balloon (Experimental): Fetal endoscopic tracheal occlusion using the Smart-TO balloon. Balloon removal procedure by peripheral course around the MR scanner
  Interventions: Other: Fetoscopic Endoluminal Tracheal Occlusion with the Smart-TO Balloon

INTERVENTIONS:
Other: Fetoscopic Endoluminal Tracheal Occlusion with the Smart-TO Balloon — Fetal Endoscopic Tracheal Occlusion using the Smart-TO balloon and non-invasive balloon removal by the peripheral magnetic field of an magnetic resonance scanner.
  Other Names: FETO

SUMMARY:
The purpose of this study is to demonstrate the ability to prenatally deflate and to evaluate the safety of the Smart-TO device for fetoscopic endoluminal tracheal occlusion (FETO) in fetuses with congenital diaphragmatic hernia and moderate to severe pulmonary hypoplasia.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) is a birth defect characterized by impaired closure of the diaphragm. This enables abdominal viscera to herniate into the thoracic cavity, leading to hypoplastic lungs and impaired lung vasculature. Fetal lung growth may be stimulated by Fetoscopic Endoluminal Tracheal Occlusion (FETO). For left-sided CDH, there is now level I evidence that it significantly improves survival in severe cases; the effect in moderate cases is much less.

Despite its benefits, the current procedure has many disadvantages. First, there is the need for prenatal reversal of the balloon, which is invasive. In utero balloon removal re-establishes airway patency. This can be done electively at 34 weeks or earlier if required, but preferentially at least 24 hours before birth. "Unplugging" requires a second procedure and a specialist team familiar with the procedure, which is available at all times. In the most extensive series published thus far, 28% of balloon removals were in an emergency setting. The only neonatal deaths were caused by complications when balloon reversal was attempted in centers without experience or unprepared. In utero reversal of the occlusion is also an invasive procedure because it requires ultrasound-guided puncture or fetoscopy. The second procedure adds both to the fetal and maternal risks.

* Balloon removal is a difficult procedure that needs expertise.
* Prenatal balloon removal procedure can fail in 3.4% even in experienced centers.
* Balloon removal is not feasible in utero in 12.6 to 24.7% of the cases.
* Balloon removal is performed in an emergency setting in 28% of the cases.
* Balloon removal can lead to neonatal death in none well-trained centers.
* In utero balloon removal may induce delivery within one week in 25% of cases.
* Patients are requested to stay close to a FETO center for the entire duration of the tracheal occlusion, which is a burden on the family, limiting the acceptability of FETO.

The Smart-TO balloon allows remotely controlled non-invasive reversal of the occlusion. Around the balloon neck, there is a metallic cylinder and inside a magnetic ball, which acts as a valve. Deflation occurs under a strong magnetic field, as generated by a clinical MRI machine. For that, it is sufficient for the pregnant woman to walk around a clinical MRI machine. The opening of the valve induces the deflation of the balloon, which is then washed out by the fluid coming out from the lungs.

The investigators have completed the translational research that proved the safety and efficacy of this balloon for FETO and want to use this medical device for the first time in humans. The purpose of this first in-woman study is to demonstrate the ability to prenatally deflate and to evaluate the safety of the Smart-TO device for FETO in fetuses with congenital diaphragmatic hernia and moderate to severe pulmonary hypoplasia. Secondary outcomes include safety parameters.

FETO with Smart-TO balloon will be performed between 27 and 31wks + 6 days depending on the severity of pulmonary hypoplasia, according to the same technique used with the balloon usually used for the FETO procedure. Reversal of the tracheal occlusion will be performed between 34 and 34wks + 6 days or earlier if necessary. In the unlikely event of a patient with imminent signs of delivery, balloon removal will be done on placental circulation or postnatally. This will ensure the patient's safety. The patient will be asked to walk around the MR scanner to open the magnetic valve and induce the deflation of the balloon. Afterwards, an ultrasound will be performed by two experienced sonographers to assess balloon deflation. In the case of deflation failure, a second and -if necessary- a third MRI exposure will be attempted following ultrasound confirmation to ensure balloon deflation. In the case of balloon failure to deflate or any doubt about deflation, an MRI with image acquisition will be performed to (1) attempt deflation and (2) assess the airway patency. In the case of failure to deflate, balloon removal will be done by fetoscopy, placental circulation, or postnatally (depending on the clinical scenario). Within 24 hours after balloon deflation:

An MRI (with image acquisition) will be performed to locate the deflated balloon and as a second safety measure to ensure the patency of the airways.

The patient will be allowed to return to her tertiary centre of preference once the airways' patency is confirmed.

Delivery does not differ from the standard care protocol for children with CDH. In the case of MRI deflation protocol, the following will be done to locate the balloon:

1. Inspection and search of any amniotic fluid, membranes, and the placenta*
2. Standard X-ray of the newborn, which is standard, to assess lungs, airways, intubation, and location of the stomach and nasogastric tube; on that the balloon may be visible, e.g., in the stomach.
3. An ultrasound of the postpartum uterus will be done to demonstrate that the uterine cavity is empty.

The follow-up and management of the newborn will be according to the standardized management protocol of the CDH EURO Consortium. Data collection will be stopped at the moment the child is discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women carrying a fetus with isolated CDH eligible for FETO, i.e. with severe or moderate hypoplasia:

  * Left sided CDH with severe (i.e. quotient of observed-to-expected- lung-to-head ratio under 25%) or moderate pulmonary hypoplasia (observed-to-expected- lung-to-head ratios of 25 to 34.9% (any liver position), or 35 to 44.9% with intrathoracic liver herniation)
  * Right sided CDH with severe pulmonary hypoplasia (quotient of observed-to-expected- lung-to-head ratio under 50%)
* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Maternal age of 18 years or older
* Single pregnancy
* Signed informed consent
* Consent to have an ultrasound of the uterus after delivery when indicated
* Postnatal management center agrees to participate

Exclusion Criteria:

Participants eligible for this Trial must not meet any of the following criteria:

* History of allergy to latex
* Contraindication to fetoscopy and FETO (maternal diseases or technical limitations making prenatal surgery hazardous or impossible)
* Premature Membrane Rupture (PROM)
* Multiple pregnancy
* Maternal age less than 18 years
* Refusal to stay close to the UZ Leuven until balloon removal
* Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
* Participation in another interventional trial with an investigational medicinal product (IMP) or device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the ability to prenatally deflate the Smart-TO balloon by the magnetic fringe field generated by an MRI scanner | Up to 34+6 weeks of pregnancy
  • Deflation rate after MRI exposure, assessed through ultrasound (US) immediately after MRI exposure

SECONDARY OUTCOMES:
Balloon expulsion from the fetal airways after deflation. | Immediately after MRI exposure
  Absence of balloon visualization with ultrasound
Rate of spontaneous deflation of the balloon. | Up to 34+6 weeks of pregnancy
  • Spontaneous balloon deflation prior to MRI exposure, as diagnosed through ultrasound. Although a rare event, this has been reported with the standard Goldbal2® balloon in 3.1%
Percentage of lung growth | Two weeks after FETO
  • Lung growth assessed by US prior to deflation, measured by change in the observed-to-expected lung-to-head-ratio (o/e LHR) before balloon insertion and two weeks after FETO
Number of adverse events related to the balloon. | From date of inclusion until date of discharge from the hospital
Balloon localisation at birth | At birth
  • Localisation of the balloon either by (1) direct visualization within the amniotic fluid, membranes or placenta, (2) postnatal chest X-ray of the newborn, and (3) ultrasound of the postpartum uterus

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No